CLINICAL TRIAL: NCT02843672
Title: Open Randomized Controlled Clinical Trial To Assess Functional Outcomes Between Two Therapeutic Options In The Surgical Treatment Of Metatarsalgia: Triple Weil Osteotomy (Two) And Distal Metatarsal Osteotomy Minimally Invasive (DMMO)
Brief Title: Operative Treatment Of Metatarsalgia: Triple Weil Osteotomy Or Distal Metatarsal Minimal Invasive Osteotomy (DMMO)?
Acronym: WeilvsDMMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manuel Cuervas-Mons (Other)
Responsible Party: Sponsor-Investigator, Manuel Cuervas-Mons, Medical Doctor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUERVASMONS
Record Dates: First submitted 2016-07-05; First posted 2016-07-26 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Metatarsalgia
Keywords: metatarsalgia; surgery; weil; MIS; percutaneous; DMMO
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TWO (Active Comparator): Patients with metatarsalgia and without response to non-operative treatment after six months, needing surgical treatment for relief of their symptoms.
  Triple´s Weil osteotomy is performed.
  Interventions: Procedure: Triple Weil´s Osteotomy
- DMMO (Active Comparator): Patients with metatarsalgia and without response to non-operative treatment after six months, needing surgical treatment for relief of their symptoms.
  Distal metatarsal minimally invasive osteotomy is performed.
  Interventions: Procedure: Distal metatarsal minimally invasive osteotomy

INTERVENTIONS:
Procedure: Triple Weil´s Osteotomy — A 10mm longitudinal incision is made with a No.15 blade in the second intermetatarsal space immediately behind the dorsal interdigital fold, parallel to the extensor tendon. An intra-articular osteotomy in the metatarsal head is performed angled 45º relative to the long axis of the metatarsal and in a dorsal-distal to proximal-plantar direction. A second osteotomy is performed perpendicular to the metatarsal shaft,.The osteotomy is fastened with a 2.0mm snap-off screw.
  Once all the osteotomies are completed, the incisions are closed with a 2/0 monofilament suture.
  Other Names: TWO
  Arms: TWO
Procedure: Distal metatarsal minimally invasive osteotomy — A 5mm longitudinal incision is made with a MIS blade No.64 in the intermetatarsal space immediately behind the dorsal interdigital fold, parallel to the extensor tendon. Under fluoroscopy vision, an extra-articular osteotomy in the metatarsal neck is performed angled 45º relative to the long axis of the metatarsal and in a dorsal-distal to proximal-plantar direction. The osteotomies scheduled preoperatively are performed, repeating the same procedure for each ray needing an osteotomy. Once all are completed, the incisions are closed with a 4/0 monofilament suture.
  Other Names: DMMO
  Arms: DMMO

SUMMARY:
INTRODUCTION

Metatarsalgia is a vague term defining a symptom instead of a specific condition. The aim of surgical treatment of metatarsalgia is to decrease the pressure under metatarsal head, shortening and / or raising the metatarsal. It has been somewhat controversial, with more than 25 different lesser metatarsal osteotomies described to date.

The Triple´s Weil osteotomy described by Maceira is the most widely used surgical treatment in open distal metatarsal surgery but nowadays, percutaneous osteotomy has proven to be a valid technique that yields results similar to open osteotomy for the treatment of metatarsalgia and other forefoot problems. It has been somewhat controversial the choice between the different operative treatments, being nowadays the triple´s Weil osteotomy (TWO) and the distal minimally invasive osteotomy (DMMO) the most popular, gaining both defenders and retractors surgeons in open and percutaneous surgery.

The purpose of this study is to compare the clinical results between two different surgical treatments: triple´s Weil osteotomy (TWO) and distal minimal invasive osteotomy (DMMO).

MATERIAL AND METHODS

The investigators design an open randomized controlled clinical trial with patients operated in the same centre.

The patients are randomized to TWO and DMMO groups. Number of osteotomies is based on the criteria of Leventen formula. In all patients the metatarsal osteotomy can be combined with different surgical procedures in presence of associated deformities: (i) SCARF osteotomy for hallux valgus (HV) deformity, (ii) flexor and extensor tenotomies with distal phalangeal percutaneous osteotomy for lesser toes deformities.

DETAILED DESCRIPTION:
INTRODUCTION

Metatarsalgia is a vague term defining a symptom instead of a specific condition. The aim of surgical treatment of metatarsalgia is to decrease the pressure under metatarsal head, shortening and / or raising the metatarsal, thus removing the overload and preserving the joint integrity. It has been somewhat controversial, with more than 25 different lesser metatarsal osteotomies described to date. The Weil osteotomy is the most widely used surgical treatment in open distal metatarsal surgery, a popularity based upon the simple technique, stable fixation, excellent union rates and predictable results.

According to the principles of traditional surgery, surgical manoeuvres requiring large incisions and aggressive techniques should be needed to effectively resolve the different pathological elements producing the deformity in order to eliminate this serious injury. These principles concerns surgeons like White, who described a modification of the distal metaphyseal osteotomy through a percutaneous approach without visualization and without internal fixation to obtain a metatarsal in optimal weight-bearing position. Percutaneous surgery of the foot, also known as minimal invasive surgery (MIS), allows interventions to be carried out through extremely small incisions without direct exposure of the surgical field under radiologic monitoring, thus causing minimal injury to adjacent tissues, and reducing the surgical trauma. Over the last few years, Foot Surgery has come to be recognised as a major Orthopaedic subspecialty, where the percutaneous surgery plays an important role. The Triple´s Weil osteotomy described by Maceira is the most widely used surgical treatment in open distal metatarsal surgery but nowadays, percutaneous osteotomy has proven to be a valid technique that yields results similar to open osteotomy for the treatment of metatarsalgia and other forefoot problems. It has been somewhat controversial the choice between the different operative treatments, being nowadays the triple´s Weil osteotomy (TWO) and the distal minimally invasive osteotomy (DMMO) the most popular, gaining both defenders and retractors surgeons in open and percutaneous surgery.

The purpose of this study is to compare the clinical results between two different surgical treatments: triple´s Weil osteotomy (TWO) and distal minimal invasive osteotomy (DMMO).

MATERIAL AND METHODS

The investigators design an open randomized controlled clinical trial with patients operated in the same centre.

The patients are randomized to TWO and DMMO groups. Number of osteotomies is based on the criteria of Leventen formula. In all patients the metatarsal osteotomy can be combined with different surgical procedures in presence of associated deformities: (i) SCARF osteotomy for hallux valgus (HV) deformity, (ii) flexor and extensor tenotomies with distal phalangeal percutaneous osteotomy for lesser toes deformities.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive adult patients with the diagnosis of mechanical metatarsalgia served in the Department of Orthopaedic Surgery and Traumatology of the investigative hospital, without non-operative treatment response after 6 months

Exclusion Criteria:

* traumatic metatarsalgia
* secondary metatarsalgia (diabetes, rheumatoid arthritis, or general diseases)
* equinus contracture
* active infection
* systematic disease (inflammatory, metabolic, neurologic or vascular) explaining symptoms, - metatarsophalangeal (MTPJ) dislocation higher than 5mm
* inability to complete postoperative management
* previous forefoot surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline American Orthopaedic Foot and Ankle Society score (AOFAS) at 3 and 12 months | Preoperative, 3 months follow-up and 12 months follow-up
  Score for pain, function and alignment
Change from Baseline Short form Health survey 36 (SF-36) at 3 and 12 months | Preoperative, 3 months follow-up and 12 months follow-up
  Score for quality of life
Change from Baseline Visual Analog Score (VAS) at 3 and 12 months | Preoperative, 3 months follow-up and 12 months follow-up
  Score for pain
Benton-Weil´s questionnaire | 12 months follow-up
  The questionnaire incorporate actual VAS and clinical results subjectively evaluated with three questions:
  (i) Does the surgery meet your expectations? (ii) Would you recommend the procedure to a friend in similar conditions? (iii) Would you have undergone the procedure, knowing now your outcome?

SECONDARY OUTCOMES:
Change from 3 months MTPJ joint mobility at 12 months | 3 months follow-up and 12 months follow-up
  Metatarso-phalangeal joint (MTPJ) mobility described as the range of motion (ROM) of the joint, measured by a goniometer MTPJ range of motion is measured in a open chain patient who is lying down with the knee extended and the foot at rest in spontaneous plantar flexion.
  Full ROM of plantar flexion combined with dorsiflexion was classified in: normal ROM ≥70º, moderately stiff ROM 30º to 70º, and severely stiff ROM < 30º..
Change from Baseline Metatarsal formula at 12 months | Preoperative and 12 months follow-up
  Changes in the radiological metatarsal formula are measured with the average recoil of the metatarsal heads between the preoperative and the 12 months follow up measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No